CLINICAL TRIAL: NCT00426296
Title: An Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of a Fixed-Dose Combination of Abacavir 600 mg/Lamivudine 300 mg Once-Daily in Combination With Atazanavir 300 mg + Ritonavir 100 mg Once-Daily in Antiretroviral-Naïve HIV-1 Infected Subjects With Continuing Evaluation of Abacavir/Lamivudine Plus Atazanavir 400 mg for Maintenance Over an Additional 48 Weeks
Brief Title: SHARE: Simple HAART With Abacavir, Reyataz, and Epivir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Alliance for Research & Education - Infectious Diseases, LLC. (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL102060
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: HIV; Reyataz; atazanavir; Norvir; ritonavir; Boosted; Lipodystrophy; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Atazanavir Sulfate; Ritonavir

INTERVENTIONS:
Drug: atazanavir (Reyataz)
Drug: ritonavir (Norvir)

SUMMARY:
SHARE: Simple HAART with Abacavir, Reyataz, and Epivir

DETAILED DESCRIPTION:
Open-label, multicenter study of ABC/3TC + ATV in subjects who have completed at least 24 weeks of treatment on ABC/3TC+ATV/RTV as their first line regimen and have plasma HIV-1 RNA <50 copies/mL at entry

ELIGIBILITY:
Inclusion Criteria:

* Currently taking abacavir/lamivudine (Epzicom) in combination with atazanavir (Reyataz) boosted with ritonavir (Norvir) as first antiretroviral regimen
* Viral load <50 copies/ml

Exclusion Criteria:

* Viral load >50 copies/ml
* Having taken more than one antiretroviral regimen

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Elion, MD, Principal Investigator — Whitman-Walker Clinic
Locations (1):
- Whitman-Walker Clinic, Washington D.C., District of Columbia, United States